CLINICAL TRIAL: NCT06305884
Title: Project Limb Rescue: A Pilot Study Evaluating the Feasibility of Transcutaneous Sensors for the Detection of Cancer-Related Lymphedema
Brief Title: Transcutaneous Sensors for the Detection of Cancer-Related Lymphedema, Project Limb Rescue Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Carlo Contreras, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSU-21287; NCI-2023-03077 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Lymphedema; Malignant Solid Neoplasm
MeSH Terms: conditions — Lymphedema | interventions — Exercise; Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (BI, PPG) (Experimental): Participants undergo BIA and wear "watch-like" sensors and undergo PPG at rest and while active (pedaling an exercise bike) on study.
  Interventions: Procedure: Bioelectric Impedance Analysis; Other: Exercise; Procedure: Photoplethysmography; Behavioral: Questionnaire Administration

INTERVENTIONS:
Procedure: Bioelectric Impedance Analysis — Undergo BI
  Other Names: BIA; Bioelectric Impedance; Bioelectric Impedance Test; Bioelectrical Impedance Analysis; Bioimpedance Analysis
Other: Exercise — Pedal an exercise bike
  Other Names: Exercise Type
Procedure: Photoplethysmography — Undergo PPG
  Other Names: PPG
Behavioral: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies how well new adhesive-based sensors that stick to the skin (transcutaneous) work in detecting cancer-related long-term arm swelling (lymphedema). For many patients, lymphedema s painful, unsightly, and weakening. The early signs of lymphedema are hard to see, and sometimes it is only diagnosed by hospital equipment at larger centers. Treating lymphedema early is usually more successful than trying to treat in later stages. The adhesive-based sensors used in this study work by using techniques called photoplethysmography (PPG) and bioimpedance (BI). PPG is an optical technique that can be used to detect blood volume changes in tissue. BI evaluates how tissue responds to an externally applied electrical current. This study may assist researchers in distinguishing participants with lymphedema in comparison to participants without lymphedema, and develop a way for patients to check for lymphedema at home.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Describe a unique signature using a combination of photoplethysmography and bioimpedance that distinguishes participants with lymphedema in comparison to participants without lymphedema at rest.

SECONDARY OBJECTIVES:

I. In participants with lymphedema, describe a unique signature using a combination of photoplethysmography and bioimpedance that distinguishes the affected arm in comparison to the unaffected arm.

II. Tolerability of the transcutaneous sensors during the participant data collection session.

III. Use a combination of photoplethysmography and bioimpedance to identify likely cut points for lymphedema in participants with lymphedema.

OUTLINE:

Participants undergo BI and wear "watch-like" sensors and undergo PPG at rest and while active (pedaling an exercise bike) on study.

ELIGIBILITY:
Inclusion Criteria:

* COHORT A: Healthy participants
* COHORT B: Participants with pre-existing lymphedema
* COHORT B: A history of cancer therapy with surgery or radiation involving the axillary basin
* COHORT B: Unilateral upper extremity swelling that requires compression or pneumatic therapy or a >= 2-centimeter difference in contralateral arm circumference

Exclusion Criteria:

* Patients with active malignancy or ongoing cancer therapy will be excluded, though breast cancer patients currently on endocrine monotherapy will be included

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Unique signature describing photoplethysmography and bioimpedance at rest and during activity | Up to 2 hours
  Will assess in the following groups: (1) Healthy dominant arm, (2) healthy recessive arm, (3) lymphedema normal arm and (4) lymphedema affected arm. A single continuous value will be developed from the amplitude over time for each participant, both at rest and during activity. These measurements will be summarized using descriptive statistics (means, standard deviations or medians and interquartile ranges).

SECONDARY OUTCOMES:
Patient reported outcomes | Up to 2 hours
  Assess by the Lymph-Q questionnaire. Will be summarized by cohort and compared between cohorts using the methods outlined above for continuous variables and either a Chi-square test or Fisher's Exact test for categorical variables.
Tolerability of sensors | Up to 2 hours
  Assess by the Tolerability questionnaire. Will be summarized by cohort and compared between cohorts using the methods outlined above for continuous variables and either a Chi-square test or Fisher's Exact test for categorical variables.
Likely classification for lymphedema | Up to 2 hours
  Will examine receiver operator characteristics using data from groups 3 and 4. Sensitivity, specificity, and area under that curve will be calculated, however these will be considered preliminary.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo M Contreras, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu